CLINICAL TRIAL: NCT04615390
Title: Recovery Profiles in Patients With COVID-19 Outcomes Undergoing Rehabilitation
Brief Title: Recovery Profiles in Patients With SARS-CoV-2 Outcomes Undergoing Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, PhD, University Hospital of Ferrara
Other Study IDs: Covid-19_rehabilitation
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Covid19_rehabilitation
Keywords: covid19; rehabilitation; mindfulness; functional recovery; psychological well-being; pain; post covid syndrome
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Early rehabilitation — The intervention is primarily focused on the recovery of mobility and functional autonomy. The treatment sessions are dependent on the patient's exercise tolerance.
Behavioral: Subacute rehabilitation — Comprehensive intensive rehabilitation in the hospital
Behavioral: Mindfulness training — The home mindfulness training consists of 2 parts: 1) explanation and reflection of the Mindfulness practice 2) formal and informal practice.
Behavioral: Personalized ambulatory training — Low-intensity walking exercises at home

SUMMARY:
COVID19 patients survivors, after discharge from hospital show reduced lung function and reduced ability to exercise. Furthermore, mental health problems including stress, anxiety and depression and a low quality of life were observed. The prospective observational study involves COVID19 patients who have needed rehabilitation at the University Hospital of Ferrara. Patients receive comprehensive rehabilitation based on their specific needs in both acute and subacute rehabilitation. At the end of hospital rehabilitation, patients are offered a program to be carried out at home for both physical and psychological problems. A range of demographic and clinical data will be collected. Patients will also undergo a battery of functional, cognitive and psychological tests at 12, 26 and 52 weeks from the infection onset. Moreover, a specific assessement (both clinical and instrumental) on the pain symptom experienced, where present, will be done.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of covid19 (WHO criteria);
* indication for respiratory and / or neuromotor rehabilitation treatment

Exclusion Criteria:

* cognitive or communication impairment precluding informed consent
* severe medical conditions
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People infected with COVID-19 and healthy subjects matched for age and sex (pain assessment).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Borg scale | At the beginning of early rehabilitation
  Rating perceived exertion on a 10-points scale in which higher values correspond to havier symptomps.
Heart rate | At the beginning of early rehabilitation
  Heart rate in sitting and standing positions.
Oxygen saturation | At the beginning of early rehabilitation
  Oxygen saturation in sitting and standing positions.
30 seconds sit-to-stand test | At the beginning of early rehabilitation
  To measure the strength of the lower limbs.
Change in 1 minute sit-to-stand test between two time points | Month 3, Month 6
  To measure the strength of the lower limbs.
Change in Short form health survey between three time points | At the beginning of early rehabilitation, Month 3, Month 6
  Is a general health questionnaire for the assessment of the patient's quality of life. Two summary scores are reported: a mental component score and a physical component score. The scores may be reported as Z-scores.
2-minute walking test | At the beginning of early rehabilitation
  For mobility assessment
Change in 6-minute walking test between two time points | Month 3, Month 6
  For mobility assessment
Change in Functional Independence Measure Scale between two time points | At the beginning of early rehabilitation, Month 3
  Evaluate the functional autonomy of the patient both on the motor and cognitive side (minumum score:18 maximum score:126 ). At 3 months the "FIM efficiency" is evaluated as a measure of the efficiency of the rehabilitation intervention.
Change in Montreal Cognitive Assessment (MoCA) between two time points | Month 3, Month 6
  Cognitive screening test. Higher scores (0-30) are related to a better performance.
Cognitive Reserve Index questionnaire | Month 3
  For measuring cognitive reserve. It comprehends a overall evaluation of the subject's cognitive status based on social and personal data. Higher scores underline major cognitive reserves.
Change in Patient Health Questionnaire-9 (PHQ-9) between two time points | Month 3, Month 6
  To identify the presence of depression and measure its severity. Score goes from 0 to 27 in which higer numbers represent worse clinical outcomes.
Change in Beck Anxiety Inventory (BAI) between two time points | Month 3, Month 6
  To measure the severity of anxiety. Higher scores (0-63) indicates more severe anxiety symptoms
Change in Connor-Davidson Resilience Scale between two time points | Month 3, Month 6
  To measure the resilience. Total score goes from 0 to 40, higher points mean greater resilience.
Change in Impact of Event Scale - Revised between two time points | Month 3, Month 6
  To measure the amount of distress that associate with a specific event. Total score varies from 0 to 88, higher scores indicate greater post-event distress.
Change in General Self Efficacy Scale between two time points | Month 3, Month 6
  To assess how much people believe they can achieve their goals, despite difficulties. Total score could be from 4 to 40, higher results show larger self efficacy perception.
Change in Pittsburgh Sleep Quality Index (PSQI) between two time points | Month 3, Month 6
  To assess sleep quality. Higher scores are related to a worse sleep quality.
Covid19 Yorkshire Rehabilitation Scale (C19-YRS) | Referred changes between 3, 6 and 12 months after the symtomps onset
  Clinical interview (qualitative evaluation) for investigating perceived outcomes after the acute phase of the pathology.
Changes on pain intensity assessed with a Numeric Rating Scale (NRS) between three time points | Month 3, Month 6, Month 12
  To estimate the amount of pain perceived through a numerical classification in which higher scores indicate greater pain intensity
Changes in Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) score between three time points | Month 3, Month 6, Month 12
  To investigate neuropathic charateristics of pain. The global score goes from 0 to 24, over 12 points it is palusible the presence of neuropathic mechanism.
Changes in Central Sensitization Inventory (CSI) score between three time points | Month 3, Month 6, Month 12
  To detect the presence of central sensitization (score between 0-100 in which higher scores suggest the presence of central sensitization)
Pressure Pain Threshold (PPT) | Month 3, Month 6, Month 12
  Changes assessed with an algometer on upper trapezius and rectus femoris bilaterally
Temporal Summation (TS) | Month 3, Month 6, Month 12
  Changes assessed with an algometer on upper trapezius and rectus femoris bilaterally
Changes in Pain Catastrophizing Scale (PCS) score between three time points | Month 3, Month 6, Month 12
  To examine the pain experience felt
Changes in Tampa Scale of Kinesiophobia (TSK) score between three time points | Month 3, Month 6, Month 12
  For detecting the pain consequences on movement and related beliefs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroscience and Rehabilitation, University Hospital of Ferrara, Ferrara, Emilia-Romagna, Italy